CLINICAL TRIAL: NCT07341789
Title: Effects of Supplementation With a New Formulation of Vitamin B12, Natural Orange Extract and a Combination of Both on Physical and Mental Performance.
Brief Title: Effects of Vitamin B12 and Natural Orange Extract, and Their Combination on Physical and Mental Performance
Acronym: MECHEPS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Javier Martínez Noguera (Other)
Responsible Party: Sponsor-Investigator, Francisco Javier Martínez Noguera, Co-Principal Investigator, Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CE092504
Record Dates: First submitted 2025-12-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Vitamin b12; Supplementation During Endurance Performance; Flavonoids; Mental Fatigue; Biomarker Feedback
Keywords: Ergogenic aids; Wingate test; Vitamin B12; Polyphenols; Performance; Natural orange extract
MeSH Terms: conditions — Mental Fatigue | interventions — Vitamin B 12; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: A triple-blind, randomized, crossover clinical trial will be conducted with three experimental groups (vitamin B12 + natural orange extract; natural orange extract; and vitamin B12) and one placebo group (microcrystalline cellulose). Acute effects will be evaluated after a loading phase (three intakes, one per day including the test day). A 7-day washout period will be implemented between interventions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The company that formulated the supplements and placebo carried out the randomization, so no one on the research team or among the sponsors knew which group each study subject belonged to. The results of the randomization were sent to our laboratory after the study was completed to determine which subjects were in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin B12 (Experimental): This group will take 1.0 mg of vitamin B12 two days before the tests and 3 hours before each test. Therefore, the supplementation will last 3 days in total.
  Interventions: Dietary Supplement: Vitamin B 12
- Natural orange extract (Experimental): This group will take 500 mg of natural orange extract two days before the tests and 3 hours before each test. Therefore, the supplementation will last 3 days in total.
  Interventions: Dietary Supplement: Natural orange extract
- Vitamin B12 + natural orange extract (Experimental): This group will take 1.0 mg of vitamin B12 + 500 mg of natural orange extract two days before the tests and 3 hours before each test. Therefore, the supplementation will last 3 days in total.
  Interventions: Combination Product: Vitamina B12 + natural orange extract
- Placebo (Placebo Comparator): This group will take 500 mg of microcrystalline cellulose two days before the tests and 3 hours before each test. Therefore, the supplementation will last 3 days in total.
  Interventions: Dietary Supplement: Microcrystalline Cellulose

INTERVENTIONS:
Dietary Supplement: Vitamin B 12 — Subjects in this group will intake 1 mg/day of vitamin B12.
  Other Names: Vitamin B12
  Arms: Vitamin B12
Dietary Supplement: Natural orange extract — Subjects in this groups will intake 500 mg/day of natural orange extract.
  Arms: Natural orange extract
Combination Product: Vitamina B12 + natural orange extract — This group will take the combination of vitamin B12 and Vitamina B12 (1 mg/day) + natural orange extract (500 mg/day).
  Arms: Vitamin B12 + natural orange extract
Dietary Supplement: Microcrystalline Cellulose — Microcrystalline cellulose was used, this molecule was selected to avoid affecting the glycemia, as it can occur with dextrose or maltodextrin.
  Arms: Placebo

SUMMARY:
The aim of this study was to determine the effects of a new formulation of vitamin B12, natural orange extract, and their combination on physical and mental performance.

DETAILED DESCRIPTION:
A triple-blind, randomized, crossover clinical trial will be conducted with three experimental phases (vitamin B12 + natural orange extract, natural orange extract, vitamin B12) and one control phase (placebo), including evaluations of the acute effect after a loading phase (three intakes, one per day including the test day).

Participants

The sample will consist of 20 well-trained male cyclists (road, MTB, or triathlon), training 3-6 sessions per week, aged between 18 and 45 years. The inclusion criteria will be:

* Healthy male (to be certified through medical examination and health analysis).
* Aged 18-45 years.
* Well-trained (3-6 training sessions per week).
* Habitual consumer of citrus fruits (orange, mandarin, lemon, or grapefruit, either whole or as juice).

Tests

* General health analysis: A general blood test (including standard biochemistry and complete blood count) will be performed during the recruitment phase.
* Medical examination: A cardiorespiratory assessment at rest will be conducted to rule out any underlying pathology.
* Specific performance-related blood analysis: Conducted at four time points (total of eight measurements): baseline during recruitment, pre- and post-test in each condition (supplement / placebo). Parameters will include: complete blood count, ferritin, CK, LDH, vitamin B12, transaminases, reticulocytes, homocysteine, C-reactive protein, IL-6, methylmalonic acid, holo-transcobalamin II, 8-OHdG (8-hydroxy-2'-deoxyguanosine), dopamine, serotonin, and Brain-Derived Neurotrophic Factor (BDNF).
* Anthropometry: Determination of body composition parameters to characterize the sample.
* Wingate test: Conducted using the standard load protocol, consisting of five maximal 30-second sprints with 3-minute recovery intervals between repetitions.
* Mental fatigue test using light-based reaction tasks: The time required to complete a light reaction sequence will be measured before and after the fatigue protocol.
* Genetic test: A saliva sample will be collected to analyze genetic profiles related to food intolerances and vitamin absorption. The objective is to identify potential explanations for interindividual differences in absorption capacity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male (to be certified through medical examination and health analysis).
* Aged 18-45 years.
* Well-trained (3-6 training sessions per week).
* Habitual consumer of citrus fruits (orange, mandarin, lemon, or grapefruit, either fresh or juiced).

Exclusion Criteria:

* Smokers or regular alcohol drinkers.
* Persons suffering from a metabolic, cardiorespiratory or digestive pathology or anomaly.

digestive system.

* People who have suffered an injury in the last 6 months that limits the performance of the study tests. of the study tests.
* People taking supplements or medication in the 2 weeks before the start of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Wingate test | Throughout study completion, an average of 4 weeks
  This test consists of 5 efforts of 30 seconds at maximum intensity with a recovery of 3 minutes on a bike. In this test the peak and average power of each effort and the total average will be evaluated. In addition, the time to maximum peak power and the fatigue index.

SECONDARY OUTCOMES:
Mental fatigue test | Throughout study completion, an average of 4 weeks
  In this test, we will measure the speed of reaction in the resolution of a sequence of lights set by the researcher before and after the end of the performance test.
Hematological Parameters | Throughout study completion, an average of 4 weeks
  A complete blood count (including red blood cell count, hemoglobin, hematocrit, and white blood cell count) will be measured from venous blood samples before and after performance tests.
Iron Status Marker | Throughout study completion, an average of 4 weeks
  Serum ferritin concentration measured as an indicator of iron status, will be measured from venous blood samples before and after performance tests.
Vitamin B12 Status - Serum Vitamin B12 | Throughout study completion, an average of 4 weeks
  Serum vitamin B12 concentration measured from venous blood samples, will be measured from venous blood samples before and after performance tests.
Functional Vitamin B12 Biomarkers | Throughout study completion, an average of 4 weeks
  Description:
  Plasma methylmalonic acid, holo-transcobalamin II, and homocysteine concentrations assessed as functional biomarkers of vitamin B12 status, will be measured from venous blood samples before and after performance tests.
Muscle Damage Markers | Throughout study completion, an average of 4 weeks
  Description:
  Serum creatine kinase (CK) and lactate dehydrogenase (LDH) concentrations measured as indicators of exercise-induced muscle damage, will be measured from venous blood samples before and after performance tests.
Hepatic Enzymes | Throughout study completion, an average of 4 weeks
  Description:
  Serum glutamic-oxaloacetic transaminase (GOT/AST) and glutamic-pyruvic transaminase (GPT/ALT) concentrations, will be measured from venous blood samples before and after performance tests.
Inflammatory Marker | Throughout study completion, an average of 4 weeks
  Description:
  Serum C-reactive protein (CRP) concentration measured as a marker of systemic inflammation, will be measured from venous blood samples before and after performance tests.
Oxidative Stress Marker | Throughout study completion, an average of 4 weeks
  Description:
  Plasma 8-hydroxy-2-deoxyguanosine (8-OHdG) concentration measured as a marker of oxidative DNA damage, will be measured from venous blood samples before and after performance tests.
Neurotransmitters | Throughout study completion, an average of 4 weeks
  Description:
  Plasma serotonin, dopamine, norepinephrine, and epinephrine concentrations measured as indicators of neuroendocrine response, will be measured from venous blood samples before and after performance tests.
Neurotrophic Factor | Throughout study completion, an average of 4 weeks
  Description:
  Serum Brain-Derived Neurotrophic Factor (BDNF) concentration, will be measured from venous blood samples before and after performance tests.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Martinez Noguera, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Research Center for High Performance Sport. Universidad Católica de Murcia, La Ñora, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No